CLINICAL TRIAL: NCT04684693
Title: Effect of Laser Puncture on Rheumatoid Arthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, A. Sedky, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/010-2020
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Experimental)
  Interventions: Device: Laser
- Control Group (Active Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Laser — Laser puncture and exercise
  Arms: Laser Group
Procedure: Control — Exercise
  Arms: Control Group

SUMMARY:
Studying the effect of laser puncture on rheumatoid arthritis patients

ELIGIBILITY:
Inclusion Criteria:

* Meeting the criteria of ACR classification for rheumatoid arthritis
* Meeting the criteria of EULAR classification for rheumatoid arthritis

Exclusion Criteria:

* Having malignancy
* Having connective tissue disease
* Smokers

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-01-22 (Estimated)

PRIMARY OUTCOMES:
HAQ (Change) | Pre-intervention, 4 weeks
  Health Assessment questionnaire
RAQoL (Change) | Pre-intervention, 4 weeks
  Rheumatoid Arthritis Quality of Life
CRP (Change) | Pre-intervention, 4 weeks
  Analysis of serum C-reactive protein
IL-6 (Change) | Pre-intervention, 4 weeks
  Plasma interleukin-6 inflammatory markers
ATP (Change) | Pre-intervention, 4 weeks
  Plasma ATP concentration anti-oxidant marker
MDA (Change) | Pre-intervention, 4 weeks
  plasma malondialdehyde oxidative marker

CONTACTS AND LOCATIONS:
Locations (1):
- M. Sedky, Cairo, Egypt

REFERENCES:
- [Derived] Adly AS, Adly AS, Adly MS, Ali MF. A novel approach utilizing laser acupuncture teletherapy for management of elderly-onset rheumatoid arthritis: A randomized clinical trial. J Telemed Telecare. 2021 Jun;27(5):298-306. doi: 10.1177/1357633X211009861. Epub 2021 May 9. PMID 33966520